CLINICAL TRIAL: NCT02697071
Title: A Randomized Placebo-Controlled Trial of Sub-Dissociative Ketamine for Treatment of Acute Migraine-Type Headache in the Emergency Department
Brief Title: Ketamine for Acute Migraine in the Emergency Department
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Carilion Clinic (Other)
Collaborators: Virginia Polytechnic Institute and State University (Other)
Responsible Party: Principal Investigator, Corey Heitz, Director of Undergraduate Medical Education, Department of Emergency Medicine, Carilion Clinic
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1921
Record Dates: First submitted 2016-02-24; First posted 2016-03-03 (Estimated); Results first posted 2021-02-25 (Actual); Last update posted 2021-03-26 (Actual); Status verified 2021-03

CONDITIONS: Headache
Keywords: Ketamine; Migraine; Headache; Emergency Department
MeSH Terms: conditions — Headache; Migraine Disorders; Emergencies | interventions — Ketamine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (2):
- Placebo Control (Placebo Comparator): Patients will receive an equivalent volume of normal saline intravenously.
  Interventions: Drug: Normal Saline
- Ketamine (Experimental): Patients will receive 0.2mg/kg ketamine intravenously over one minute.
  Interventions: Drug: Ketamine

INTERVENTIONS:
Drug: Ketamine — Patients in this arm will receive 0.2mg/kg ketamine intravenously, pain scores will be collected after 30 minutes. At that time rescue medication will also be offered. Pain scores will continued to be recorded until 60 minutes have passed since drug administration.
  Arms: Ketamine
Drug: Normal Saline — Patients will receive normal saline intravenously, pain scores will be collected after 30 minutes. At that time rescue medication will also be offered. Pain scores will continued to be recorded until 60 minutes have passed since drug administration.
  Arms: Placebo Control

SUMMARY:
This research study will be a prospective, randomized, double-blind, placebo-controlled trial. Because ketamine has yet to be directly studied as treatment for acute migraine headache in the emergency department, the research team is initially interested if ketamine can reduce pain scores in headache patients and reduce the incidence of recurrence while exhibiting an adequate safety profile. By using a placebo-controlled study design, the research team can adequately investigate the effectiveness of the medication in a subgroup previously not well studied.

DETAILED DESCRIPTION:
The investigators propose enrollment of patients upon or shortly after presentation to the emergency department for treatment with ketamine or placebo. 30 minutes after study drug is administered, patients will have the option to request rescue medication which will be ordered by the treating physician according to standard emergency department protocol. Pain scores will be documented using the Numerical rating scale (NRS-11), 4-Point Pain Intensity Categorical Scale, and 4-Point Functional Disability Scale at 0 minutes, 30 minutes, and 60 minutes post treatment. Follow-up telephone calls will be made 72-120 hours after treatment to assess the incidence of recurrence of head pain and patient satisfaction with the treatment.

Subjects eligible for this study must present to the emergency department with a chief complaint of primary headache that is determined non-emergent by the treating physician.

Upon block randomization, each subject will receive an intravenous dose of 0.2 mg/kg, with a maximum dose of 30mg, of ketamine or an equivalent volume of saline. After 30 minutes patients will be asked if they need rescue medication, and the treating physician will administer rescue treatment, if requested.

The research hypotheses include:

1. The proportion of patients achieving significant pain reduction at 30 minutes will be higher in the ketamine treatment group compared to the placebo group.
2. The proportion of patients experiencing pain response, defined as <50% reduction in the visual analog score compare to the baseline and a reduction of the 4-Point Pain Intensity Categorical Scale to a 1 or 0, will be higher for patients receiving ketamine compared to those receiving the placebo.
3. Patients treated with ketamine for headache will experience lower recurrence rates within 24 hours
4. Ketamine will demonstrate an adequate safety profile.

The last two questions will be exploratory and not included in the power analysis.

It is expected that ketamine will demonstrate a satisfactory safety profile with limited side effects. The proportion of patients attaining pain response is expected to be higher in the ketamine treatment group compared to placebo. It is also expected that patients treated with ketamine alone will be less likely to experience a recurring headache within 72 hours of treatment than those treated with placebo and rescue medication.

The primary outcome will be achievement of pain response at 30 minutes after ketamine dose. Achievement of pain response will be defined as reduction in baseline pain score by at least 50% on the NRS scale. Secondary outcomes will include attainment of pain-free state, patient headache relief, recurrence of headache, recovery of functional disability, and need for rescue medication.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years of age
* Chief complaint of headache
* International Classification of Headache Disorder classification of migraine or probable migraine with or without aura
* Has decision making capacity
* Consent
* Provider determination of non-emergent cause

Exclusion Criteria:

* Over the age of 50 with first time headache
* Known adverse reaction or tolerance to study medication
* Headache due to trauma
* New onset, focal, abnormal, neurologic findings
* New onset seizures
* History of metastatic cancer or neoplasm
* Active psychotic symptoms
* Altered mental status
* Provider intends to preform lumbar puncture
* Pregnancy
* Breast feeding
* Previous enrollment in study
* Fever > 100.3 F
* Physiologic instability (blood pressure < 90/50 or >170/100, heart rate <50 or >120, chronic respiratory, renal or hepatic failure)
* Suspected cardiac pain

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2016-02; Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Corey Corey, MD, Principal Investigator — Carilion Clinic
Locations (1):
- Carilion Roanoke Memorial Emergency Department, Roanoke, Virginia, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo Control | Ketamine
Started | 18 | 16
Completed | 18 | 16
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo Control | Ketamine | Total
Number analyzed (Participants) | 18 | 16 | 34
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.5 (8.3) | 38.5 (13.75) | 34.3 (11.75)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 13 | 26
  Male | 5 | 3 | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 3 | 5
  White | 13 | 10 | 23
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 3 | 3 | 6
Region of Enrollment [Number; unit: participants]
  United States | 18 | 16 | 34
Headache duration [Count of Participants; unit: Participants]
  Days (>24h) | 6 | 5 | 11
  Hours (<24h) | 11 | 10 | 21
  Weeks (>7d) | 1 | 1 | 2
Self-medicated before ED presentation [Count of Participants; unit: Participants] | 15 | 13 | 28
Visual Aura Present [Count of Participants; unit: Participants] | 6 | 5 | 11
International Classification of Headache Disorders [Count of Participants; unit: Participants] — Participants were categorized using the International Classification of Headache Disorders (ICD-3) into groups based on migraine without (1.1) or with aura (1.2), or probably migraine without (1.5.1) or with (1.5.2) aura. https://ichd-3.org/1-migraine/
  Participants
    1.1 - Migraine without aura | 9 | 8 | 17
    1.2 - Migraine with aura | 3 | 5 | 8
    1.5.1 - Probably migraine without aura | 3 | 2 | 5
    1.5.2 - probably migraine with aura | 3 | 1 | 4
Baseline categorical pain intensity [Count of Participants; unit: Participants]
  Severe | 12 | 14 | 26
  Severe-moderate | 1 | 0 | 1
  Moderate | 4 | 2 | 6
  Mild | 1 | 0 | 1
Baseline functional disability [Count of Participants; unit: Participants]
  No disruption | 0 | 0 | 0
  Mildly impaired | 5 | 4 | 9
  Moderately impaired | 6 | 6 | 12
  Severely impaired | 7 | 6 | 13
Baseline NRS [Median (Inter-Quartile Range); unit: scores on a scale] — NRS = numerical rating scale for pain, from 0-10, where 0 is no pain, and 10 is the most pain they have felt/can imagine feeling. 1-3 are "mild", 4-6 are "moderate", and 7-10 are considered "severe" pain.
  scores on a scale | 8 [7 to 9] | 8.25 [7.75 to 10] | 8 [7 to 9.75]

OUTCOME MEASURES:

1. Primary Outcome: Achievement of Pain Response After Ketamine Dose.
Description: NRS (National rating scale) pain score change from baseline following ketamine dose. Minimum score is 0, maximum score is 10, and higher scores mean worse pain.
Time Frame: 30 minutes
Measure: Median (Inter-Quartile Range); unit: change in score on a scale
Arm/Group | Placebo Control | Ketamine
Number analyzed (Participants) | 18 | 16
change in score on a scale | 2.0 [0 to 3.75] | 1.0 [0 to 2.25]

2. Secondary Outcome: Categorical Pain Score Change From Baseline
Description: change in baseline categorical pain score at 30 minutes (categorical pain intensity score from 0 to 3 where 0="no headache" and 3="severe headache")
Time Frame: 30 minutes
Measure: Mean (95% Confidence Interval); unit: change in score on a scale
Arm/Group | Placebo Control | Ketamine
Number analyzed (Participants) | 18 | 16
change in score on a scale | 0.72 [0.61 to 0.83] | 0.56 [0.44 to 0.68]

3. Other Pre Specified Outcome: Functional Disability Score Change From Baseline
Description: change in functional disability from baseline at 30 minutes (functional disability score from 0 to 3 where 0="no disruption of daily activities" and 3="performance of daily activities is severely impaired")
Time Frame: 30 minutes
Measure: Mean (95% Confidence Interval); unit: change in score on a scale
Arm/Group | Placebo Control | Ketamine
Number analyzed (Participants) | 18 | 16
change in score on a scale | 0.39 [0.3 to 0.48] | 0.44 [0.32 to 0.56]

ADVERSE EVENTS:
Time Frame: 1 month
Arm/Group | Placebo Control | Ketamine
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/16
Other Adverse Events (participants affected / at risk) | 0/18 | 0/16

LIMITATIONS AND CAVEATS:
A limitation in our study was the chosen ketamine dose. The subjective quality of patient-reported data in pain studies is a limitation.

Another limitation in our study was maintaining strict control over additional medications given before or within 30 minutes of study drug administration.

Another limitation was quantification of worsening migraine side effects. The final limitations include study location and sample size - single institution in a small city surrounded by a rural area.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-06-06): https://cdn.clinicaltrials.gov/large-docs/71/NCT02697071/Prot_SAP_000.pdf